CLINICAL TRIAL: NCT03809715
Title: Post-marketing Clinical Follow-up Study With Coroflex® ISAR Neo
Brief Title: Coroflex ISAR NEO "All Comers" Post Market Clinical Follow-up (PMCF)
Status: Completed | Type: Observational
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1803
Record Dates: First submitted 2019-01-17; First posted 2019-01-18 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Coroflex® ISAR NEO coronary stent system — treatment of coronary artery disease with Coroflex® ISAR NEO of "real world" de-novo and restenotic lesions in native coronary arteries and coronary bypass grafts

SUMMARY:
The aim of the study is to assess the safety and efficacy of the device to treat coronary de novo and restenotic lesions.

DETAILED DESCRIPTION:
Post-authorisation / after Conformité Européene (CE) marking Coroflex® ISAR NEO is a drug eluting stent system which is an improved version of the predecessor device Coroflex® ISAR which was extensively studied in the ISAR 2000 Registry. The rationale of this observational, post-market, single-armed study is to confirm the safety and efficacy of Coroflex® ISAR NEO, also as part of the manufacturer's post-market surveillance obligations in particular for the re-certification of the device.

ELIGIBILITY:
Inclusion Criteria:

Coroflex® ISAR NEO is intended to be used for

* All common significant coronary lesions
* Target lesion length >34mm need to be covered with at least 2 stents
* Patients eligible for this study must be at least 18 years of age.
* The patient must fulfill the standard recommendations for Percutaneous Coronary Intervention (PCI) based on the last European Society of Cardiology (ESC) recommendations within his/ her regular treatment or that the use of the product has already been decided within the regular planning of the patient's treatment.

Exclusion Criteria:

* Intolerance to sirolimus and/or probucol
* Allergy to components of the coating
* Pregnancy and lactation
* Complete occlusion of the treatment vessel because of an unsuccessfully re-canalized
* Cardiogenic shock
* Risk of an intraluminal thrombus
* Hemorrhagic diathesis or another disorder such as gastro-intestinal ulceration or cerebral circulatory disorders which restrict the use of platelet aggregation inhibitor therapy and anti-coagulation therapy
* Surgery shortly after myocardial infarction with indications of thrombus or poor coronary flow behavior
* Severe allergy to contrast media
* Lesions which are untreatable with PCI or other interventional techniques
* Patients with an ejection fraction of < 30 %
* Vascular reference diameter < 2.00 mm
* Treatment of the left stem (first section of the left coronary artery)
* Indication for a bypass surgery
* Contraindication for whichever accompanying medication is necessary

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The investigator of each study site has the responsibility of screening all potential patients and selecting those who fulfil the inclusion criteria of this study protocol. Therefore, at each site a study with similar inclusion criteria cannot be conducted while the recruitment of this study is in progress.
  Screening will be performed during the physical examination to verify the "patient related enrolment criteria". The second part of the screening procedure will be completed during the diagnostic angiography to verify that the target lesion fulfils all "lesion related enrolment criteria".
Sampling Method: Non-Probability Sample
Enrollment: 3520 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Target Lesion Revascularization (TLR) rate at 12 months | 12 months

SECONDARY OUTCOMES:
Accumulated Major Adverse Cardiovascular Events (MACE) rate at 12 months (including intra-hospital events) | 12 months
  MACE consists of all events TLR (Re-Percutaneous Coronary Intervention (Re-PCI), Coronary Artery Bypass Grafting (CABG)), Myocardial Infarction (MI), cardiac death (inhospital) and all-cause death up to 12 months. MI is defined as a new event documented with elevated cardiac enzymes during the follow-up. Elevated enzyme levels during the hospital stay are not considered as a new event.
Accumulated Target Vessel Failure Rate at 12 months (including intra-hospital events) | 12 months
Stent thrombosis rates accumulated up to 12 months | 12 months
  Stent thrombosis is defined as thrombosis in the treated coronary lesion only. No venous thrombotic events are relevant for this end point.
Rate of bleeding complications accumulated up to 12 months | 12 months
  To assess the bleeding complications the Bleeding Academic Research Consortium (BARC) scale will be used.
Technical/procedural success rate | immediately after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Rene Koning, MD, Principal Investigator — Clinique St. Hilaire
Locations (1):
- Clinique St. Hilaire, Rouen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Landolff Q, Quillot M, Picard F, Henry P, Sideris G, Bizeau O, Piot C, Jouve B, Rischner J, Mejri M, Charmasson C, Lasserre R, Pouliquen H, Joseph T, Monsegu J, Karsenty B, Martin Yuste V, Richet N, Lapeyre G, Beverelli F, Beygui F, Koning R. In-Hospital and 1-Year Clinical Results from the French Registry Using Polymer-Free Sirolimus-Eluting Stents in Acute Coronary Syndrome and Stable Coronary Artery Disease. J Interv Cardiol. 2023 Dec 13;2023:8907315. doi: 10.1155/2023/8907315. eCollection 2023. PMID 38125031